CLINICAL TRIAL: NCT05732480
Title: Understanding Changes in the Gut Microbiome in Patients With Gallstone Disease and Its Impact on Patient Outcomes
Brief Title: Influence of Gut Microbiome in Gallstone Disease
Status: Recruiting | Type: Observational
Sponsor: East Kent Hospitals University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2022/SURG/01
Record Dates: First submitted 2023-02-07; First posted 2023-02-17 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Gall Stone; Gall Stones, Common Bile Duct; Pancreatitis; Acute Cholecystitis
MeSH Terms: conditions — Gallstones; Pancreatitis; Cholecystitis, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — We are collecting stool samples to analyse bacterial DNA however patient DNA will also be present in these samples. Samples will be destroyed at the end of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this prospective observational study is to explore the role of the gut microbiome in patients with gallstone disease.

The main question[s] it aims to answer are:

* if there is a relationship between the gut microbiome and the development of complications associated with gallstone disease (such as pancreatitis and acute cholecystitis)
* if there are changes in the gut microbiome following cholecystectomy and the relationship with patient outcomes.

Participants will be asked to provide stool samples at fixed time points (recruitment, pre- and post-cholecystectomy if applicable and at 6 months and 3 years. They will also be asked to provide stool samples if they represent to hospital with complications associated with their gallstone disease.

DETAILED DESCRIPTION:
Background:

Gallstone disease affects 10-15% of people in the United Kingdom (UK) and over 65,000 patients undergoing cholecystectomy each year, costing the National Health Service (NHS) over 110 million. There is increasing evidence suggesting differences in the gut microbiome of patients with gallstone disease compared to those without (including reduced diversity, decreased prevalence of beneficial and increased prevalence of pathogenic bacteria) but there are only a handful of small scale studies exploring the development of gallstone disease complications and patient outcomes to date.

Hypothesis and Objectives:

This pilot study aims to understand the profile of the gut microbiome in adult patients diagnosed with gallstone disease and its relationship with patient outcomes including:

Patients who develop complications of gallstone disease(including but not limited to biliary colic, cholangitis, cholecystitis, pancreatitis and gallstone ileus) following diagnosis and Patients who develop post-operative complications including short (hospital stay, wound healing etc) and intermediate (development of post-cholecystectomy diarrhoea) outcomes.

Design and Methods:

A prospective cohort design will be used to collect data from 75 adult patients presenting to East Kent University Hospitals NHS Foundation Trust Hospitals with newly diagnosed gallstone disease following confirmatory imaging investigations.

Data will be collected from electronic patient records including clinical history and diagnostic investigations, anthropometry, blood and imaging results (if taken as part of routine clinical care) for the initial presentation and subsequent readmissions/planned follow-up timepoints.

Stool samples will be collected from patients either during admission or at home at each timepoint. Samples will be returned by post to the research team where they will be stored and analysed. Patients will also be asked to provide a 3 day food diary card Patients will have a sample collected at time of diagnosis and then at 6 monthly intervals whilst awaiting cholecystectomy. A pre-operative sample will be required within 6 weeks of any surgical intervention. Following cholecystectomy an immediate post-operative sample (within the first week) will be collected as well as a sample at 6 months.

Clinical and Scientific Impact:

At least 20% of those patients awaiting cholecystectomy experience complications, costing the NHS over £25 million per year. Therefore, there is a huge need to understand mechanisms behind the development of complications and to reduce the symptom burden for patients as well as the financial burden for the NHS.

This study is the crucial first step in identifying differences in the gut microbiome between patients who experience complications (both pre and post-op) and those who do not. Once differences are discovered the next step will be to use the information discovered to determine interventions to reduce the development of these complications.

ELIGIBILITY:
Inclusion Criteria:

* All adults (age >18 years of age) patients diagnosed with gallstone disease following confirmatory imaging at an East Kent University Foundation Trust Hospital. Patients of any gender, ethnicity or socio-economic background are eligible as well as pregnant women. Patients undergoing both open and laparoscopic cholecystectomy will be included.

Exclusion Criteria:

* Patients less than 18 years of age and patients who do not have capacity to consent to involvement in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with gallstone disease presenting to an East Kent University Foundation Trust Hospital
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2023-05-30 (Actual); Primary Completion 2025-11-13 (Estimated); Study Completion 2026-11-13 (Estimated)

PRIMARY OUTCOMES:
Bacterial DNA profile | through study completion, up to 3 years from cholecystectomy
  The diversity of species present in the stool of participants

CONTACTS AND LOCATIONS:
Locations (1):
- EKHUFT, Ashford, Kent, United Kingdom